CLINICAL TRIAL: NCT00108459
Title: Safety and Efficacy of Low Carbohydrate Diet in Obesity and Type 2 DM: RCT
Brief Title: Low Carbohydrate Diet Compared to Calorie and Fat Restricted Diet in Patients With Obesity and Type II Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDA-002-03F
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-07

CONDITIONS: Obesity; Type 2 Diabetes; Hyperlipidemia
Keywords: Obesity; Type 2 Diabetes; Hyperlipidemia; Insulin resistance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Hyperlipidemias; Insulin Resistance | interventions — Diet, Carbohydrate-Restricted

INTERVENTIONS:
Behavioral: Low Carbohydrate Diet

SUMMARY:
This study is designed to address the hypothesis that in obese patients with type 2 diabetes mellitus (DM), a low carbohydrate diet not specifically restricted in calories compared to low fat, caloric restricted diet over 24 months will cause 5% greater reduction in body weight in patients with obesity and type 2 DM, be safe, and will not have any detrimental effects on serum lipid concentrations.

DETAILED DESCRIPTION:
Objectives:

This study is designed to address the hypothesis that in obese patients with type 2 DM, a low carbohydrate diet not specifically restricted in calories compared to low fat, caloric restricted diet over a 24 months period will:

* Primary:

  1. Cause 5% greater reduction in body weight in patients with obesity and type 2 DM;
  2. Be safe and will not have any detrimental effects on serum lipid concentrations
* Secondary:

  1. Lead to a greater reduction in HbA1c and fasting serum glucose and insulin concentration;
  2. Lead to reduction in body fat content;
  3. Cause greater reduction in serum triglyceride concentration;
  4. Cause no significant changes in proteinuria, serum low-density lipoprotein (LDL), high-density lipoprotein (HDL), creatinine and uric acid concentrations
* Exploratory:

Cause favorable changes in adipocytokines (serum leptin, resistin, TNF-α, TNF α- receptors, free fatty acids) and high sensitive C-reactive protein

Research Design:

This will be a single site (Philadelphia VA Medical Center); two arm, parallel, randomized, clinical trial. Obese, male, type 2 diabetic subjects (body mass index [BMI] >30 kg/m2) will be randomized in a 1:1 fashion to dietary instructions for low carbohydrate or low fat diet. Women will be randomized separately (blocks of 4) to ensure equal representation in both dietary groups. Recruitment will be done in 3 phases (for logistical reasons). Subjects will be randomized to one of the two dietary groups. One group will be instructed on a carbohydrate-restricted diet, and the other on a calorie and fat restricted diet as recommended by the National Heart, Lung and Blood Institute (NHLBI). All patients will have blood, urine, and body composition analyses measured at baseline and then at 26, 52, and 104 weeks. Dietary instructions will be given to subjects in groups of 13, and will be provided every week for the first 4 weeks and then every 4 weeks for a total of 30 visits.

Methodology: The setting is the outpatient clinics of the Philadelphia Veterans Affairs Medical Center. Inclusion criteria include: Male or female subjects > 18 years of age; Clinical diagnosis of type 2 diabetes mellitus; Body mass index of > 30 kg/m2 . Approximately 156 male and female veterans from the Philadelphia Veterans Affairs Medical Center will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 18 years of age
* Clinical diagnosis of type 2 diabetes mellitus or on insulin or oral hypoglycemic agents
* Body mass index of > 30 kg/m2
* The subject must we willing and able to monitor their blood glucose with a glucometer at least 2 times per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2004-09; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Nayyar Iqbal, Principal Investigator — VA Research
Locations (1):
- VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Iqbal N, Vetter ML, Moore RH, Chittams JL, Dalton-Bakes CV, Dowd M, Williams-Smith C, Cardillo S, Wadden TA. Effects of a low-intensity intervention that prescribed a low-carbohydrate vs. a low-fat diet in obese, diabetic participants. Obesity (Silver Spring). 2010 Sep;18(9):1733-8. doi: 10.1038/oby.2009.460. Epub 2009 Dec 17. PMID 20019677